CLINICAL TRIAL: NCT01833663
Title: Multi-site, Randomized, Opened and Controlled Comparison Study on the Effectiveness and Safety of Solifenacin Succinate Tablets and Solifenacin Succinate Tablets + Estrogen for Overactive Bladder in the Post-menopausal Women
Brief Title: Effectiveness and Safety Study of Solifenacin Succinate and Solifenacin Succinate + Estrogen to Treat OAB in Postmenopausal Women
Acronym: OAB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Astellas Pharma China, Inc. (Industry); Beijing CAT Science Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XH-WXK-001
Record Dates: First submitted 2013-04-10; First posted 2013-04-17 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Overactive Bladder; Postmenopausal Disorder; Urination Disorders
Keywords: Overactive Bladder; Solifenacin Succinate Tablets; Estrogen
MeSH Terms: conditions — Urinary Bladder, Overactive; Urination Disorders | interventions — Solifenacin Succinate; Estrogens

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Solifenacin Succinate Tablets and Estrogen capsules (Experimental): Solifenacin Succinate Tablets (5mg/d) + local estrogen for 12 weeks
  Interventions: Drug: Solifenacin Succinate Tablets; Drug: Estrogen
- Solifenacin Succinate Tablets (Active Comparator): Solifenacin Succinate Tablets (5mg/d) for 12 weeks
  Interventions: Drug: Solifenacin Succinate Tablets

INTERVENTIONS:
Drug: Solifenacin Succinate Tablets
Drug: Estrogen
  Arms: Solifenacin Succinate Tablets and Estrogen capsules

SUMMARY:
This study is a multi-site, randomized, opened and parallel-controlled clinical study.

The patients up to the inclusion criteria are randomly treated with Solifenacin Succinate Tablets (5mg/d) or Solifenacin Succinate Tablets (5mg/d) + local estrogen for 12 weeks. Before the dosing and at Week 4, 8 and 12 of the dosing, various examinations are made, and various indices are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women aged ≤75.
* Signing of ICF.
* Willing to and able to correctly complete the urination diary.
* Complications of OAB for ≥12 weeks (including: urgent micturition, frequent urination (≥8 times in the daytime, and ≥2 times at the night) and/or urgent urinary incontinence).
* No dosing of other drugs of same kind within 14d. -≥8 urination times (24h) in the 1d urination diary.

Exclusion Criteria:

* Clinically-significant dysuria(at the investigators' viewpoints).
* Serious stress urinary incontinence or mixed stress/urgent urinary incontinence (mainly stress one) confirmed by the investigators.
* At the ongoing intubatton or the intermittent self-intubatton.
* Evidence-based urinary tract infection or chronic inflammation in the recent 2 weeks (e.g. interstitial cystitis), bladder calculus, past pelvic radiotherapy, and past or existing pelvic malignant tumors.
* Uncontrolled narrow-angle glaucoma, urinary/gastric retention, intestinal obstruction and other medical symptoms forbidden for anti-cholinergic drugs at the investigators' viewpoints.
* Non-pharmacotherapy (including electrotherapy) or bladder training within 2 weeks before the study initiation (or during the study).
* Dosing of diuretics and drugs with the cholinergic or anti-cholinergic adverse reactions
* Known or suspicious allergy to Solifenacin Succinate, other anti-cholinergic drugs or lactose.
* Clinically-significant symptoms inapplicable for clinical study at the investigators' viewpoints.
* Participation in other clinical studies within 30d before the random grouping.
* No completion of urination diary according to relevant instructions.
* Potentially clinically significant abnormalities (PCSA) inapplicable for clinical study at the investigators' viewpoints.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Difference between the mean urination times (24h) at the end of treatment and the baseline value | 12 weeks

SECONDARY OUTCOMES:
Difference between the mean urgent micturition times (24h) and the baseline value | on week 12

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhu, doctor, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401